CLINICAL TRIAL: NCT03193749
Title: A Trial Testing Amiodarone in Chagas Cardiomyopathy (ATTACH)
Brief Title: A Trial Testing Amiodarone in Chagas Cardiomiopathy
Acronym: ATTACH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Collaborators: Instituto de Corazón de Bucaramanga (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 880-2015; 277872553480 (Other Grant/Funding Number: Colciencias)
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Chagas Cardiomyopathy
Keywords: Chagas disease, cardiomyopathy, amiodarone, clinical trial
MeSH Terms: conditions — Chagas Cardiomyopathy; Chagas Disease; Cardiomyopathies | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amiodarone Hydrochloride (Experimental): Oral treatment for at least 6 months
  Interventions: Drug: Amiodarone Hydrochloride
- Placebo (Placebo Comparator): Oral treatment for at least 6 months
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Amiodarone Hydrochloride — Starting (loading) dose 400 mg PO once a day for 10 days. Maintainance dose 200 mg PO once a day for at least 6 months, up to 24 months
  Arms: Amiodarone Hydrochloride
Drug: Placebo Oral Tablet — Matching placebo for tablets of 200 mg of Amiodarone
  Arms: Placebo

SUMMARY:
Purpose:

The ATTACH trial, as currently designed, will primarily test whether a treatment with Amiodarone for at least 6 months has a trypanocidal effect among individuals with mild-to-moderate Chronic Chagas Cardiomyopathy. A secondary goal will be to confirm, in this population, a clinical benefit from this treatment (in terms of reducing mortality or cardiac arrhythmic events), and to explore whether a potential trypanocidal effect is associated with a clinical benefit.

DETAILED DESCRIPTION:
Investigators currently plan to enroll over 200 participants in Bogotá and Bucaramanga, Colombia. Such sample size will provide 82% of statistical power to detect at least a 30% relative reduction in the primary outcome. This is assuming that at least 75% of untreated participants will test positive at least once after three qualitative PCR assays for Trypanosoma cruzi during the 6th month after randomization (allowing for up to 10% losses to follow up and treatment adherence over 90%).

ATTACH is currently seeking collaborating centers internationally. The current funding structure will allow to test study hypothesis on trypanocidal effect, whereas data on clinical effects will be exploratory. Investigators expect to increase the sample size to at least 600 participants in order to a) enhance geographical variability/generalizability for the primary results and b) to achieve enough statistical power to test the hypothesis on clinical impact.

New centers are welcome to join this protocol, either as a placebo-controlled or as a pragmatic, open label trial. These centers will be working with the central coordination with their own funding/logistic capabilities. In the open label protocol, eligible, consenting participants will be randomly prescribed or not to Amiodarone. As assessing clinical impact will be the priority, new centers are not required to have on-site PCR capabilities. These centers are encouraged to store blood samples for PCR testing elsewhere later, if possible.

See details on eligibility, interventions and outcome measures below

ELIGIBILITY:
ATTACH will enroll individuals with positive serology for Trypanozoma cruzi and evidence of both structrural and rythm/conduction cardiac abnormalities, as defined by any of the following inclusion criteria

1. Structural cardiac abnormality (at least one):

   * NTpro-BNP values >125 ng/ml, or BNP values > 50 ng/ml
   * Left ventricular ejection fraction (LVEF) <50% or left diastolic diameter > 5.5 cm
   * Symptoms of heart failure, or one episode of acute heart failure over the last 12 months
2. Rrythm/conduction cardiac abnormality (at least one)

   * EKG monitoring showing 10 or more VPBs/hour or ventricular Tachycardia
   * EKG showing left anterior hemiblockade or right bundle branch blocakde
   * Use of a cardiac stimulation device as treatment for A-V block or Sinus node dysfunction

The protocol allows concurrent treatments for the condition (e.g. beta-blockers, ACE inhibitors, etc.) other than Amiodarone. Individuals meeting the above eligibility criteria who have previously received trypanocidal therapy (e.g. Benznidazole or Nifurtimox) can still be included, as long as they prove to be PCR positive for T. cruzi at enrollment. Co-intervention with these agents during the study will also be allowed, as per physician's judgment, either as open label treatment, or as part of another study not involving Amiodarone.

Exclusion criteria:

* LVEF < 30% or NYHA Class III-IV
* Medical prescription with chronic use of Amiodarone
* Pregancy (currently, or planned in the following 2 years), or childbearing age without reliable birth control
* Heart rate < 50 or AV blockade without treatment with cardiac stimulation device
* Contraindication for Amiodarone as per treating physician (e.g. because of long QT syndrome, thyroid disease, interstitial lung disease)
* Atrial fibrillation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Positive PCR for Trypanosoma cruzi | 6 months after starting treatment
  Conventional (qualitative) Polymerase Chain Reaction. At least one positive result out of three tests at least one week apart from each other

SECONDARY OUTCOMES:
Composite of clinical events | Up to study closure or 24 months after randomization (whichever comes first)
  a) All-cause deaths; b) EKG-supported ventricular tachycardia or, c) Hospitalization for cardiac causes
Elements of the composite outcome of clinical events individually | Up to study closure or 24 months after randomization (whichever comes first)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Villar, MD, MSc, PhD, Principal Investigator — Department of Research, Fundación Cardioinfantil - Instituto de Cardiología; Diego A Rodriguez, MD, Principal Investigator — Department of Cardiology, Fundación Cardioinfantil - Instituto de Cardiología
Locations (1):
- Fundación Cardioinfantil - Instituto de Cardiología, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Upon submission of primary results, following requests of editors, by request to the steering committee

REFERENCES:
- [Background] Rassi A Jr, Rassi A, Little WC, Xavier SS, Rassi SG, Rassi AG, Rassi GG, Hasslocher-Moreno A, Sousa AS, Scanavacca MI. Development and validation of a risk score for predicting death in Chagas' heart disease. N Engl J Med. 2006 Aug 24;355(8):799-808. doi: 10.1056/NEJMoa053241. PMID 16928995
- [Background] Rassi A Jr, Rassi A, Rassi SG. Predictors of mortality in chronic Chagas disease: a systematic review of observational studies. Circulation. 2007 Mar 6;115(9):1101-8. doi: 10.1161/CIRCULATIONAHA.106.627265. PMID 17339568
- [Background] Veiga-Santos P, Barrias ES, Santos JF, de Barros Moreira TL, de Carvalho TM, Urbina JA, de Souza W. Effects of amiodarone and posaconazole on the growth and ultrastructure of Trypanosoma cruzi. Int J Antimicrob Agents. 2012 Jul;40(1):61-71. doi: 10.1016/j.ijantimicag.2012.03.009. Epub 2012 May 14. PMID 22591838
- [Background] Adesse D, Azzam EM, Meirelles Mde N, Urbina JA, Garzoni LR. Amiodarone inhibits Trypanosoma cruzi infection and promotes cardiac cell recovery with gap junction and cytoskeleton reassembly in vitro. Antimicrob Agents Chemother. 2011 Jan;55(1):203-10. doi: 10.1128/AAC.01129-10. Epub 2010 Nov 15. PMID 21078932
- [Background] Benaim G, Sanders JM, Garcia-Marchan Y, Colina C, Lira R, Caldera AR, Payares G, Sanoja C, Burgos JM, Leon-Rossell A, Concepcion JL, Schijman AG, Levin M, Oldfield E, Urbina JA. Amiodarone has intrinsic anti-Trypanosoma cruzi activity and acts synergistically with posaconazole. J Med Chem. 2006 Feb 9;49(3):892-9. doi: 10.1021/jm050691f. PMID 16451055